CLINICAL TRIAL: NCT06796699
Title: A Multi-center, Single-Arm, Open-Label Phase Ia/Ib Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of GH56 Capsules in Subjects With MTAP-Deleted Advanced Solid Tumors
Brief Title: A Phase Ia/Ib Clinical Study of GH56 Capsules in Subjects With MTAP-Deleted Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH56C101
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors With MTAP Gene Deletion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GH56 Capsule Group (Experimental): Participants will be randomized to receive one of 6 active dose levels of GH56 orally (PO) daily (QD) in 21 days cycles. The study will determine the recommended dose of expansion (RDEs) and RP2D.
  Interventions: Drug: GH56 Capsule

INTERVENTIONS:
Drug: GH56 Capsule — GH56 capsule for oral administration at specified doses on scheduled days.

SUMMARY:
This is a multicenter, single-arm, open-label, dose-escalation, dose-expansion study to evaluate the safety, tolerability, PK/PD, and preliminary anti-tumor activity of GH56 Capsule in subjects with advanced solid tumors who have failed or are intolerant in standard treatment, or have no standard therapy. The clinical trial will be carried out in two parts: phase Ia study (dose escalation study) and phase Ib (dose expansion study).

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing to participate in the clinical trial, understand and sign the informed consent, and comply with the study visits and procedures.
* 2. Men or women ≥18 years old.
* 3. Men or women with MTAP-Deleted Advanced Solid Tumors.
* 4. Subjects with solid tumors must have at least one evaluable lesion which should be measurable by RECIST v1.1.
* 5. Eastern Cooperative Oncology Group (ECOG) performance status (Table 12) 0 to 1.
* 6. Survival expectations ≥ 12 weeks.
* 7. Subjects with adequate organ function and the laboratory test critera.
* 8. Serum pregnancy test (for female of childbearing potential) negative within 7 days prior to first dosing of study treatment. Male and female subjects of childbearing potential must agree to use effective methods of contraception from the time of ICF signed, throughout the study and for 6 months after the last dose of the investigational product. A patient is of childbearing potential if, in the opinion of the Investigator, he/she is biologically capable of having children and is sexually active.

Exclusion Criteria:

* 1. Subject has not recovered from a prior surgical procedure or has undergone any major surgery within 4 weeks prior to the first dose.
* 2. Known (including suspected) allergic to GH56 or its components.
* 3. Has received any anti-tumor agents within 28 days without delayed toxicity for the treatment of advanced tumors prior to the first administration of GH56 Capsule or has received radiation therapy, biologic therapy, endocrine therapy, targeted therapy, immunotherapy, or other anti-tumor drug treatments within 28 days prior to the first administration of GH56 Capsule, or other anti-tumor drugs or treatments within the following interval before the first administration of GH56 Capsule.
* 4. Has symptomatic or active progressive central nervous system (CNS) metastases such as molluscum contagiosum metastases.
* 5. Subjects who have difficulty in swallowing and have a history of gastrointestinal surgery or other relevant medical disorders that may interfere with the absorption of GH56.
* 6. Subjects had a malignant tumor other than the current tumor within 5 years prior to the first administration of GH56 Capsule, except for localized cancers that have been apparently cured or without disease progression or recurrence for at least 5 consecutive years.
* 7. Uncontrolled or significant cardiovascular disease
* 8. Subjects with documented positive virology status of hepatitis, as confirmed by Screening hepatitis B virus (HBV) and hepatitis C virus (HCV) tests, Human Immunodeficiency Virus (HIV).
* 9. Conditions that the investigator considers inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
1. Determination of Maximum Tolerated Dose (MTD) , RDEs of GH56. | Approximately 3 years
  MTD is the highest dose of a treatment that does not cause unacceptable side effects.
  RDEs stand for Recommended Dose for Expansion.
Characterize the Safety of GH56 | Approximately 3 years
  Number of participants with treatment-emergent adverse events and serious AEs.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Disease Control Rate (DCR) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Progression-Free Survival (PFS) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Cmax | Approximately 3 years
  The maximum or "peak" concentration of GH56 observed after administration
Tmax | Approximately 3 years
  The time to peak concentration of GH56
T1/2 | Approximately 3 years
  Half-life of GH56
PD of GH56 | Approximately 3 years
  Change of sDMA protein expression in tumor tissues

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai GoBroad Caner Hospital China Pharmaceutical University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi